CLINICAL TRIAL: NCT01707966
Title: Orteronel Maintenance Therapy in Patients With Metastatic Castration Resistant Prostate Cancer and Non-progressive Disease After First-line Docetaxel Therapy: a Multicenter Randomized Double-blind Placebo-controlled Phase III Trial.
Brief Title: Orteronel Maintenance Therapy in Patients With Metastatic Castration Resistant Prostate Cancer and Non-progressive Disease After First-line Docetaxel Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAKK 08/11; 2011-002965-39 (EudraCT Number)
Record Dates: First submitted 2012-09-13; First posted 2012-10-16 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; metastatic castration-resistant prostate cancer; maintenance therapy; orteronel; TAK-700
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orteronel and best supportive care (Experimental): Arm A: 300mg Orteronel twice daily and best supportive care until occurrence of an event.
  Interventions: Drug: Orteronel
- Placebo and best supportive care (Placebo Comparator): Arm B: Placebo twice daily and best supportive care until occurrence of an event.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orteronel
  Other Names: TAK-700
  Arms: Orteronel and best supportive care
Drug: Placebo
  Arms: Placebo and best supportive care

SUMMARY:
The main objective of this multicenter, randomized, double-blind, placebo-controlled phase III trial is to assess the impact of maintenance orteronel on disease progression and hence on quality of life in patients with metastatic castration-resistant prostate cancer who have achieved at lease disease stabilization after first line chemotherapy with docetaxel.

DETAILED DESCRIPTION:
Background:

One in six men will be diagnosed with cancer of the prostate during his lifetime. Accordingly, prostate cancer is the most common cancer amongst men in the western world. In Switzerland approximately 5'400 men are diagnosed with the disease and 1'300 die of prostate cancer every year. Prostate cancer represents 30% of all cancer diagnoses in men. Despite earlier detection and new treatments the life time risk to die of prostate cancer has remained stable at 3% since 1980.

Metastatic prostate cancer is hormone-sensitive and therefore androgen deprivation therapy (ADT) is the treatment of choice. Yet, virtually all patients with metastatic prostate cancer progress on androgen deprivation therapy (so called castration-resistant prostate cancer: CRPC). Further hormonal manipulations are often administered (e.g. maximal androgen blockade with addition of a non-steroidal antiandrogen such as bicalutamide), however these interventions have only modest impact. Metastatic CRPC (mCRPC) that progresses despite these therapies is nowadays treated with docetaxel-based chemotherapy. In a phase III trial, treatment of mCRPC patients with docetaxel in combination with low dose prednisone resulted in a significant survival advantage in comparison to the previous standard of care of mitoxantrone plus prednisone. Moreover docetaxel treatment improved response rate, progression free survival and symptom control.

The current standard of care in patients with disease stabilization after first line chemotherapy with docetaxel is a wait-and-watch strategy, where patients are regularly examined in the hospital every 3-4 weeks. A second line chemotherapy in patients with mCRPC was not standardized until recently. However, two trials presented in 2010 have changed the landscape: the novel taxane cabazitaxel was tested in a phase III trial against mitoxantrone as a second line chemotherapy in patients progressing under or after docetaxel. There was a significant improvement in overall survival, progression free survival and response rate. Most of the included patients had experienced disease progression during or within three months of docetaxel first line treatment. Cabazitaxel was associated with increased toxicity including 5% toxic deaths. Another randomized phase III trial using abiraterone in patients with progression after docetaxel showed a significant improvement in overall survival and pain palliation. Abiraterone belongs to a group of agents that very effectively inhibits the androgen synthesis via blockade of the key enzyme cytochrome P-450c17 (CYP17).

The new drug orteronel (TAK-700) belongs to the same group of active substances as abiraterone. Orteronel is currently the subject of a large international Phase III study in patients with metastatic carcinoma of the prostate and progression of disease following docetaxel. Initial results have shown that orteronel effectively inhibits testosterone synthesis and, in contrast to abiraterone, has fewer side effects.

Rational:

CYP17 inhibitors are active and well tolerated agents for treatment of patients with castration-resistant prostate cancer. However, despite its activity patients become resistant to this new form of antihormonal treatment and hence develop further progression after a median of approximately 6 months. In that case, the options are very limited as outlined above.

In all reported post-docetaxel trials and in the large phase III trials, patients start on the CYP17 inhibitor treatment at the time of disease progression. Trials examining other advanced malignant diseases such as lung cancer have shown that initiating an effective treatment earlier in the disease course at the end of a first-line chemotherapy (so called switch maintenance therapy) is beneficial in terms of progression free survival (PFS) but also overall survival (OS). This may also hold true for early administration of antihormonal agents in patients with mCRPC.

Therefore, the aim of this trial is to test the hypothesis that starting orteronel after disease stabilization with docetaxel prolongs event-free survival (EFS), consequently maintains a good quality of life (QL) and eventually also improves OS.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given voluntary written informed consent
* Male patient 18 years or older
* WHO performance status of ≤2
* Adenocarcinoma of the prostate
* Castration resistance: tumor progression after orchiectomy or during treatment with GnRH analogues
* Metastatic disease, radiographically documented (
* Total testosterone ≤ 50 ng/dL
* Non-progressive disease after docetaxel first-line treatment with a cumulative dose ≥ 300mg/m2

  * No evidence of progression on imaging according to PCWG2 and modified RECIST 1.1 criteria
  * PSA levels not elevated ≥ 25% AND at least 2 ng/mL above the nadir since start of docetaxel treatment
* Non-surgically castrated patient agrees on ongoing use of GnRH analogues (agonists or antagonists) during the trial
* PSA ≥ 2 ng/mL; Potassium ≥ 3.5 mmol/L; Neutrophils ≥ 1.5 x 109/L; Platelets ≥ 100 x 10x9/L
* Normal kidney and liver function
* Planned start of trial treatment 3 to 6 weeks after last docetaxel administration
* Screening calculated ejection fraction of ≥ 50% or normal according to local standard by echocardiogram or by multiple gated acquisition (MUGA) scan.
* Baseline QL questionnaire completed
* Patient is able and willing to swallow study drug as whole tablet
* Patient compliance and geographic proximity allow proper staging and follow-up
* Patient agrees to practice effective barrier contraception or to completely abstain from intercourse

Exclusion Criteria:

* Prior therapy with aminoglutethimide, ketoconazole, orteronel, abiraterone or other modern CYP17 inhibitors
* Prior chemotherapy for prostate cancer within 12 months before enrollment except from docetaxel
* Retreatment with docetaxel after interruption of > 5 weeks
* Concurrent disease requiring higher doses of corticosteroid than the equivalent of 10 mg prednisone per day
* Known hypersensitivity to trial drug or hypersensitivity to any of its components
* Patient has received other investigational drugs within 30 days before enrollment
* Presence of a small cell component in histological specimen
* Radiotherapy within the last 2 weeks before expected start of the trial treatment
* Known history of central nervous system (CNS) or spinal cord metastases
* Current spinal cord compression
* Diagnosed or treated for another malignancy within 2 years of registration, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, or any in situ malignancies
* History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade ≥ 3 (NCI CTCAE version 4.0) or thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events) within 6 months prior to first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed
* New York Heart Association Class III or IV heart failure
* ECG abnormalities of:

  * Q-wave infarction, unless identified ≥ 6 months prior to registration
  * QTc interval > 460 msec
* Uncontrolled hypertension despite appropriate medical therapy
* Likely inability (e.g. due to a psychiatric disorder) to understand information on trial related topics, to give informed consent, to comply with the protocol, to fill in QL forms and to cooperate fully with the investigator and site personnel
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of orteronel
* Known active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Event free survival (EFS) | At baseline; every 4 weeks until disease progression (estimated up to 1 year)

SECONDARY OUTCOMES:
Adverse events (AEs) | Throughout treatment phase (estimated up to 1 year) until 30 days after last drug administration or prior to start of subsequent anticancer treatment (whichever occurs first)
Prostate-specific antigen (PSA) response (30%, 50%, 90% and best) | PSA level at baseline and every 4 weeks until disease progression (estimated up to 1 year)
Time to PSA progression | PSA level at baseline and every 4 weeks until disease progression (estimated up to 1 year)
Radiographic progression-free survival (rPFS) | Every 12 weeks until disease progression (estimated up to 1 year)
QL and pain response | First 6 months of trial treatment
Overall survival (OS) | time from trial randomization to the date of death from any cause (estimated up to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cathomas, MD, Study Chair — Kantonsspital Graubünden; Silke Gillessen, Prof, Study Chair — Cantonal Hospital of St. Gallen
Locations (15):
- Switzerland (15):
  - Kantonspital Aarau, Aarau
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Freiburg, Fribourg
  - Hôpitaux Universitaires de Genève HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Spital Männedorf, Männedorf
  - Kantonsspital Muensterlingen, Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cathomas R, Crabb SJ, Mark M, Winterhalder R, Rothermundt C, Elliott T, von Burg P, Kenner H, Hayoz S, Vilei SB, Rauch D, Roggero E, Mohaupt MG, Bernhard J, Manetsch G, Gillessen S; Swiss Group for Clinical Cancer Research SAKK. Orteronel Switch Maintenance Therapy in Metastatic Castration Resistant Prostate Cancer After First-Line Docetaxel: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial (SAKK 08/11). Prostate. 2016 Dec;76(16):1519-1527. doi: 10.1002/pros.23236. Epub 2016 Jul 25. PMID 27457964